CLINICAL TRIAL: NCT04103580
Title: Caregiver Speaks: A Technologically Mediated Storytelling Intervention for Family Caregivers of Individuals With Alzheimer's Disease and Other Dementias
Brief Title: Caregiver Speaks: A Technologically Mediated Storytelling Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Debra Parker Oliver, Professor, Division of Palliative Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016062 R01AG59818-01A1
Record Dates: First submitted 2019-07-25; First posted 2019-09-25 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Randomized 2 arm study; control and intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Will receive usual hospice care plus measures
- Intervention (Experimental): Will receive photo elicitation intervention and will join a secret Facebook group to share photos with other caregivers
  Interventions: Behavioral: Photo elicitation

INTERVENTIONS:
Behavioral: Photo elicitation — Caregivers are taught to use photos to illustrate various feelings and meanings
  Arms: Intervention

SUMMARY:
Caregiver speaks is a randomized trial of a Photo elicitation intervention for caregivers of Alzheimers patients.

DETAILED DESCRIPTION:
This randomized controlled trial will test an intervention for an understudied population - family caregivers of persons living with dementia (PLWD). This project is the first of its kind to longitudinally follow family caregivers of PLWD into bereavement. Furthermore, the intervention, Caregiver Speaks, employs an innovative storytelling approach - photo elicitation (the use of photos to elicit thoughts, feelings, and reactions to a person's experience) - to encourage family caregivers to make meaning of their caregiving and bereavement experiences as a way of reducing depression, anxiety, and ultimately grief intensity. Caregiver Speaks is deployed via a readily available social media network (Facebook), which allows easy access for already overburdened family caregivers of PLWD, and can improve their social support. Preliminary work demonstrates that 1) this project is feasible as an RCT intervention study of caregiver experiences, 2) the research team can conduct this type of storytelling intervention via Facebook, and 3) family caregivers use (and want to use) social media during active caregiving and into bereavement, despite their heavy care burdens. The research team will base the proposal on Park and Folkman's meaning-making model of stress and coping. This model illustrates how individuals cope with adverse life events (i.e., trauma, or death of a loved one) by reconstructing and transforming the event's meaning and incorporating the reappraised meaning into one's larger self-narrative. Caregiver Speaks uses storytelling in the form of photo-elicitation, in order to facilitate this meaning-making. Caregivers share photos and discussions regarding their caregiving and bereavement experiences in a private, facilitated Facebook group. This model suggests that caregivers' ability to make sense of (meaning making), and find benefit in an adverse life situation (caregiving and bereavement) will be validated through social support, and result in reduced depression, anxiety, and grief intensity. Caregivers will be randomly assigned to either: 1) Group 1, which will receive the Caregiver Speaks intervention, or 2) Group 2, which will receive standard care, including the standard care for bereavement. The research team will use both quantitative and qualitative methods in parallel and equal status to measure the intervention's efficacy. The overall hypothesis is that participating in Caregiver Speaks during caregiving and into bereavement will reduce caregivers' depression and anxiety, and as a result will reduce grief intensity in bereavement. The three specific aims are to: 1) determine the efficacy of the Caregiver Speaks intervention in reducing depression and anxiety among family caregivers of people with dementia, 2) examine the intervention's effect on grief intensity among bereaved family caregivers of people with dementia, and 3) describe how caregivers made meaning of their caregiving and bereavement experiences.

ELIGIBILITY:
Inclusion Criteria:

1. be a designated family caregiver (i.e., a family member or friend providing unpaid care) of a PLWD who is enrolled in hospice care,
2. be at least 18 years old,
3. be involved in decisions related to their loved one's hospice care,
4. have access to a digital camera or other photo-taking device such as a cell phone
5. be willing to photograph images they feel capture their caregiving and bereavement experiences
6. be willing to set up a Facebook account and join the private Facebook group, 7) have access to e-mail for REDCap survey data collection

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Parker Oliver, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment considered complete and random assignment made only after the baseline survey was completed. The baseline analysis population excludes those who were not truly randomized. Some participants who cared for the same patient were assigned to the same group (without any randomization) as the first participant from that cohort who was truly randomized. These are recorded as "Not truly randomized" as a category of participants under "Incomplete" in each phase.
Period: Phase 1 Active Caregiving
Arm/Group | Control | Intervention
Started (A participant is considered started if they completed the baseline survey.) | 227 | 230
Completed (A participant is considered completed if they completed at least one follow-up in active caregiving.) | 144 | 113
Not Completed | 83 | 117
Not completed — Lost to Follow-up | 18 | 45
Not completed — Withdrawal by Subject | 5 | 14
Not completed — Decertified from Hospice | 3 | 1
Not completed — Care Recipient Died before First Follow-up | 41 | 35
Not completed — Not truly randomized (cohort-randomized with other family caregivers) | 13 | 19
Not completed — Other | 3 | 3
Period: Phase 2 Bereavement
Arm/Group | Control | Intervention
Started (A participant is considered started in Phase 2 if they completed the first measure after patient died. Note that some participants who completed a follow-up in Phase 1 may have chosen not to continue into Phase 2 which results in the number of completed in Phase 1 to not match the number of started in Phase 2.) | 134 | 85
Completed (A participant is considered completed in Phase 2 if they completed at least one follow-up measure in bereavement.) | 117 | 62
Not Completed | 17 | 23
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Not truly randomized (cohort-randomized with other family caregivers) | 6 | 7
Not completed — Other | 8 | 6

BASELINE CHARACTERISTICS:
Population: The baseline analysis population excludes those who were not truly randomized. Some participants who cared for the same patient were assigned to the same group (without any randomization) as the first participant from that cohort who was truly randomized, so these additional participants were not included in our analysis since we do not consider them truly randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 214 | 211 | 425
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 7 Participants were missing age data.
  years
    number analyzed (Participants) | 212 | 206 | 418
    (all) | 60.2 (11.0) | 60.7 (9.69) | 60.5 (10.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 176 | 174 | 350
  Sex: Male | 36 | 37 | 73
  Sex: Other | 1 | 0 | 1
  Sex: Unknown | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 207 | 196 | 403
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 39 | 36 | 75
  White | 166 | 162 | 328
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 4 | 8 | 12
GAD-7 [Mean (Standard Deviation); unit: units on a scale] — Measure for depression measured by 7 items with 0-3 ratings. Total scores range from 0-21. Higher means greater depressive symptoms. Population: 25 participants were missing data on at least 1 item required to calculate a total GAD-7 score.
  units on a scale
    number analyzed (Participants) | 204 | 196 | 400
    (all) | 8.33 (5.92) | 8.41 (5.29) | 8.37 (5.61)
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Measure for depression measured by 9 items with 0-3 ratings. Total scores range from 0-27. Higher means greater depressive symptoms. Population: 28 participants were missing data on at least one of the items required to calculated a total PHQ-9 score.
  units on a scale
    number analyzed (Participants) | 198 | 199 | 397
    (all) | 7.20 (6.39) | 7.31 (5.63) | 7.25 (6.01)

OUTCOME MEASURES:

1. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7) Anxiety Score
Description: Caregiver anxiety measure. Response options range from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 21. Higher scores indicate more anxiety.
Time Frame: Data were collected at baseline, 14, 30, 90, 150 days in active caregiving phase and 14, 30, 90, 150, and 180 days in bereavement phase. Follow-up data were included in the calculation of score change per day as long as participant had 1 followup.
Population: Each analysis population includes participants that had at least one follow-up after first measure in each phase.
Measure: Least Squares Mean (Standard Error); unit: score on a scale change per day
Groups:
- Control - Phase 1: Control group in active caregiving
- Intervention - Phase 1: Intervention group in active caregiving
- Control - Phase 2: Control group in bereavement
- Intervention - Phase 2: Intervention group in bereavement
Arm/Group | Control - Phase 1 | Intervention - Phase 1 | Control - Phase 2 | Intervention - Phase 2
Number analyzed (Participants) | 137 | 108 | 112 | 61
score on a scale change per day | -0.014 (0.003) | -0.008 (0.004) | -0.005 (0.002) | -0.013 (0.003)
Statistical Analysis 1: Comparison: Control - Phase 1 vs Intervention - Phase 1; The null hypothesis is that there is no difference between control and intervention over time in Phase 1; Test type: Superiority; p = 0.247, Mixed Models Analysis; Due to uneven space between time points (days), we estimated a random effects model with varying intercepts and slopes for each phase independently; Slope = 0.005, Standard Error of Mean 0.005 — We used an interaction between time and study arm to determine whether there was a significant difference over time in the change in outcome. The estimate is the difference in change over time for the intervention group compared to the control group
Statistical Analysis 2: Comparison: Control - Phase 2 vs Intervention - Phase 2; The null hypothesis is that there is no difference between control and intervention over time in Phase 2; Test type: Superiority; p = 0.049, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = -0.008, Standard Error of Mean 0.004 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Patient Health Questionnaire-9 (PHQ-9) Depression Score
Description: Caregiver depression measure. Response options range from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27. Higher scores indicate more depression.
Time Frame: as for outcome 1
Population: Each analysis population includes participants that had at least one follow-up after first measure in each phase.
Measure: Least Squares Mean (Standard Error); unit: score on a scale change per day
Arm/Group | Control - Phase 1 | Intervention - Phase 1 | Control - Phase 2 | Intervention - Phase 2
Number analyzed (Participants) | 131 | 105 | 112 | 61
score on a scale change per day | -0.007 (0.003) | -0.001 (0.003) | -0.011 (0.002) | -0.013 (0.003)
Statistical Analysis 1: Comparison: Control - Phase 1 vs Intervention - Phase 1; The null hypothesis is that there is no difference between control and intervention over time in Phase 1; Test type: Superiority; p = 0.150, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = 0.006, Standard Error of Mean 0.004 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Control - Phase 2 vs Intervention - Phase 2; The null hypothesis is that there is no difference between control and intervention over time in Phase 2; Test type: Superiority; p = 0.635, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = -0.002, Standard Error of Mean 0.004 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline through 150 days in the active caregiving phase, and first measure after patient death through 180 days in the bereaved phase. Events were monitored while participants was enrolled in the study, which in some cases was shorter than the duration of assessment (150 days in active caregiving phase/180 days in bereavement phase).
Description: This is a minimal risk study and thus it is unlikely a serious adverse event would occur due to the nature of the intervention.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/230
Serious Adverse Events (participants affected / at risk) | 0/227 | 0/230
Other Adverse Events (participants affected / at risk) | 0/227 | 0/230

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04103580/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT04103580/SAP_001.pdf